CLINICAL TRIAL: NCT06719726
Title: Evaluating Preoperative PECS I Block and Intraoperative Local Anesthetic Infiltration for Postoperative Pain in Breast Augmentation: A Prospective, Double-Blind, Split-Body Study
Brief Title: PECS I Block vs. Local Infiltration in Breast Augmentation Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University Hospital (Other)
Responsible Party: Principal Investigator, Mert Ersan, Asst. Prof., Yeditepe University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KAEK-21/1031
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Breast Augmentation; Pain Management in Postoperative Care; Pain Management After Surgery; Pain Management
Keywords: breast augmentation; local infiltration; PECS 1 block; pectoral nerve block; postoperative pain management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: This study utilized a Crossover design with a split-body approach, where each participant served as their own control. The intervention involved two pain management techniques:
  PECS I block: Administered to the right breast by an anesthesiologist before surgery.
  Local anesthetic infiltration: Performed on the left breast by the plastic surgeon during surgery.
  This design allowed for direct comparison of the efficacy of the two interventions (PECS I block vs. local anesthetic infiltration) in managing postoperative pain within the same participant.
  The crossover and split-body methodology minimized inter-individual variability and provided robust data on the relative effectiveness of each technique, as all other surgical and anesthetic factors were standardized across both sides.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PECS I Block Intervention Arm (Experimental): This arm involves the application of a preoperative PECS I block with 10 mL of 0.5% bupivacaine under ultrasound guidance. The intervention targets the right breast, aiming to evaluate its effectiveness in managing postoperative pain compared to local anesthetic infiltration.
  Interventions: Procedure: PECS I Block
- Local Anesthetic Infiltration Intervention Arm (Experimental): This arm involves the administration of intraoperative local anesthetic infiltration using 10 mL of 0.5% bupivacaine under direct visualization. The intervention targets the left breast, aiming to compare its effectiveness in managing postoperative pain against the PECS I block.
  Interventions: Procedure: Local Anesthetic Infiltration

INTERVENTIONS:
Procedure: PECS I Block — The PECS I block is a regional anesthesia technique performed preoperatively under ultrasound guidance. It involves the injection of 10 mL of 0.5% bupivacaine between the pectoralis major and pectoralis minor muscles to block the medial and lateral pectoral nerves. This procedure targets the right breast in the study to reduce postoperative pain and is compared to local anesthetic infiltration.
  Arms: PECS I Block Intervention Arm
Procedure: Local Anesthetic Infiltration — Local anesthetic infiltration involves the intraoperative administration of 10 mL of 0.5% bupivacaine under direct visualization into the pectoralis major muscle prior to muscle transection. This procedure targets the left breast in the study for pain management and is compared to the PECS I block.
  Arms: Local Anesthetic Infiltration Intervention Arm

SUMMARY:
This study aimed to compare the effectiveness of preoperative PECS I block and intraoperative local anesthetic infiltration in managing postoperative pain following breast augmentation surgery. The primary focus was to evaluate their impact on postoperative pain levels, perioperative remifentanil and postoperative opioid consumption and opioid-related side effects during the early recovery period.

DETAILED DESCRIPTION:
Breast augmentation is one of the most performed procedures in aesthetic surgery worldwide.These techniques, which involve muscle dissection and manipulation, tend to be more painful compared to subglandular and subfascial placements. Thus, managing postoperative pain effectively becomes a critical aspect of patient recovery and satisfaction.

To address postoperative pain in breast augmentation, various techniques, including regional anesthesia such as pectoral nerve blocks, local anesthetic infiltration, and pocket irrigation, are employed.

This study aimed to compare the effectiveness of preoperative PECS I block and intraoperative local anesthetic infiltration in managing postoperative pain following breast augmentation surgery. The primary focus was to evaluate their impact on postoperative pain levels, perioperative remifentanil and postoperative opioid consumption and opioid-related side effects during the early recovery period.

This prospective, double-blind, split-body design study was conducted at Yeditepe University Faculty of Medicine, Plastic, Reconstructive, and Aesthetic Surgery Department, in collaboration with the Anesthesiology and Reanimation Department.

The anesthesia induction and PECS I blocks for the right breasts were performed by the same anesthesiologist in all patients (O.K.). Breast augmentation surgeries and local anesthetic infiltrations for the left breasts were performed by the same plastic surgeon (M.E.). Postoperative pain assessments were conducted by a different anesthesiologist who was blinded to the study design.

Postoperative pain was assessed using the Numeric Rating Scale (NRS), ranging from "0 = no pain" to "10 = unbearable pain." Pain assessments were performed every 30 minutes for the first 2 hours, every 2 hours between 2 and 6 hours, and at the 24ᵗʰ hour postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18 to 59 years.
* ASA (American Society of Anesthesiologists) physical status I or II.
* Scheduled for primary breast augmentation surgery using a dual-plane or submuscular approach.
* Planned to receive silicone implants of identical volume and shape for both breasts.
* Able to provide written informed consent.
* Willing and able to comply with study procedures and follow-up assessments.

Exclusion Criteria:

* Planned subglandular or subfascial breast augmentation.
* Undergoing revision breast surgery.
* History of breast disease, previous breast or axillary surgery, or breast cancer.
* Preoperative breast pain or chronic pain syndromes (e.g., fibromyalgia, chronic headaches, back pain, complex regional pain syndrome, neuropathic pain, osteoarthritis, or radicular pain).
* BIRADS score > 3 based on imaging (ultrasound/mammography) within the past year.
* Allergy to medications used in the study (e.g., bupivacaine, propofol, fentanyl, sevoflurane, cefazolin, paracetamol, ondansetron, tramadol, or morphine HCl).
* Coagulopathy or bleeding disorders.
* Pregnant or at risk of pregnancy.
* Inability to provide informed consent or communication difficulties.
* Significant medical conditions that may interfere with the study outcomes.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participation in this study is limited to self-identified women who are biologically female (cisgender women). Individuals whose self-identified gender does not align with their biological sex (e.g., transgender men, transgender women, or nonbinary individuals) are not eligible for this study. This criterion ensures consistency in evaluating outcomes related to breast augmentation surgery in a biologically female population.
Enrollment: 20 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Intensity | Up to 6 hours post-surgery.
  The level of postoperative pain in each breast region (right vs. left) measured using the Numeric Rating Scale (NRS). Pain scores will be recorded at specific intervals: every 30 minutes for the first 2 hours, every 2 hours from 2 to 6 hours, at the 24th hour, on the 5th postoperative day, and at the 3rd month. The primary focus is the pain intensity within the first 6 hours postoperatively.

SECONDARY OUTCOMES:
Opioid Consumption | Up to 24 hours post-surgery.
  Total tramadol consumption recorded within the first 6 hours and the first 24 hours postoperatively. This includes the amount administered via patient-controlled analgesia (PCA) and any additional doses required.
Opioid-Related Side Effects | Up to 24 hours post-surgery
  Incidence of opioid-related side effects such as nausea, vomiting, constipation, and respiratory depression. These will be monitored and recorded for each participant during the postoperative hospital stay
Chronic Pain Assessment | At 3 months post-surgery
  Presence of chronic pain in the breast region assessed using the Numeric Rating Scale (NRS) at the 3rd-month follow-up
Postoperative Complications | Up to 3 months post-surgery
  Incidence of complications such as wound dehiscence, hematoma, infection, implant rupture, or sensory changes in the nipple. All complications will be recorded during routine follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Mert Ersan, Asst.Prof., Principal Investigator — Yeditepe University
Locations (1):
- Yeditepe University Kozyatagi Hospital, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The following specific individual participant data (IPD) will be shared:
  De-identified Participant Data:
  Demographic data (age, BMI, ASA classification). Pain scores measured using the Numeric Rating Scale (NRS) at predefined intervals.
  Postoperative opioid consumption (tramadol and morphine requirements). Incidence of postoperative complications (e.g., sensory changes, wound dehiscence).
  Data Dictionary:
  A comprehensive guide explaining the variables and coding used in the dataset to ensure accurate interpretation by other researchers.
  Exclusions:
  Personally identifiable information (e.g., names, contact information) will not be shared to maintain participant confidentiality.
  The data will be shared after the study is completed, analyzed, and the results are published in a peer-reviewed journal. Access will be granted only to researchers who provide a justified request and agree to the terms of a formal data-sharing agreement
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data and supporting information will be made available after the study is completed, analyzed, and the results are published in a peer-reviewed journal.
  IPD and supporting documents will be shared through a secure online repository or data-sharing platform, accessible only to approved researchers
Access Criteria: Researchers must submit a formal data-sharing request, including a detailed explanation of how the data will be used.
  A data-sharing agreement must be signed to ensure the ethical use of the shared information, adherence to confidentiality, and compliance with relevant regulations.